CLINICAL TRIAL: NCT04063930
Title: A Randomized, Double-blind, Placebo Controlled, Parallel, Multicenter Study of the Effects of 12-weeks of Sodium Zirconium Cyclosilicate (Lokelma) on Albuminuria (UACR) in Patients With Type 2 Diabetes and Hyperkalemia
Brief Title: The Effect of Sodium Zirconium Cyclosilicate on Albuminuria in Patients With Type 2 Diabetes and Hyperkalemia
Acronym: ZIRCUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: AstraZeneca (Industry); Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-000595-42
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes Mellitus With Kidney Complications
Keywords: Hyperkalemia; Renin angiotensin system
MeSH Terms: conditions — Hyperkalemia | interventions — Suspensions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lokelma (Active Comparator): Sodium zirconium cyclosilicate Lokelma® 5 g, powder (Astra Zeneca)
  After initial dosing subjects will be instructed to take the study drug once daily in the morning, by oral administration after the powder has been dissolved in a glass of drinking water.
  Duration: 12 weeks
  Interventions: Drug: LOKELMA 5 GM Powder for Oral Suspension
- Placebo (Placebo Comparator): Matching placebo (indistinguishable from the active comparator)
  After initial dosing subjects will be instructed to take the study drug once daily in the morning, by oral administration after the powder has been dissolved in a glass of drinking water.
  Duration: 12 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: LOKELMA 5 GM Powder for Oral Suspension — Sodium zirconium cyclosilicate (a hyperkalemia treatment)
  Arms: Lokelma
Drug: Placebos — Matching placebo
  Arms: Placebo

SUMMARY:
To investigate whether concomitant treatment with Lokelma can improve the efficacy of standard blockade of the renin-angiotensin system in patients with type 2 diabetes, diabetic nephropathy and hyperkalemia.

DETAILED DESCRIPTION:
Patients with type 2 diabetes and nephropathy, especially patients with impaired kidney function, frequently encounter hyperkalemia as an adverse effect of RAAS blocking treatment. Consequently, RAAS blocking treatment is reduced or discontinued, which in turn impairs prognosis in terms of long-term renal and cardiovascular outcome. Not only can hyperkalemia as an adverse event lead to changes in RAAS blocking treatment, the presence of persistent potassium levels in the upper part of the normal range can impair the efficacy of the RAAS blocking treatment, another reason to expect a beneficial effect of Lokelma treatment.

The study is a multicentre (3 sites in Sweden (TBD), 2 sites in Denmark (Steno Diabetes Center Copenhagen and Zealand University Hospital, Roskilde), double-blind, randomized placebo-controlled, parallel study. The study drug is compared to matching placebo that cannot be distinguished from active drug. The treatment period is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and/or male patients with type 2 diabetes aged 18-85 years
3. Persistent macroalbuminuria (UACR ≥ 200 mg/g in at least two out of the three latest UACR measurements in subject history).
4. Chronic (at least 1 month) stable RAAS blocking treatment, i.e maximum tolerated (individually defined by investigator) dose of an ACE inhibitor or ARB at time of inclusion.
5. Documented hyperkalemia (plasma potassium ≥ 5.0 mmol/l) at least once in the 90 days prior to inclusion in the study.
6. Negative pregnancy test (urine or serum) for female subjects of childbearing potential.
7. Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of Lokelma/matching placebo to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Use of potassium-lowering agent (loop-diuretics not included)
4. Participation in another clinical study with an investigational product during the last 3 months prior to inclusion.
5. Plasma potassium < 3.5 mmol/l within the previous six months before inclusion.
6. Known hypersensitivity to Lokelma
7. Known history of drug or alcohol abuse within 1 year of screening
8. Estimated glomerular filtration rate (eGFR) <15 ml/min/1.73 m2 (calculated by CKD-EPI formula).
9. History of long QT syndrome.
10. For women only - currently pregnant (confirmed with positive pregnancy test) or breast feeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin creatinine ratio (UACR) | 12 weeks
  Change in the geometric mean of UACR (milligram per gram) measured in three consecutive morning spot urine collections from baseline to end of treatment

SECONDARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | 12 weeks
  Change in eGFR mL/min/1.73 m2 (CKD-EPI formula) from baseline to end of treatment
Urinary sodium | 12 weeks
  Change in urinary sodium levels (mmol per liter) in one 24h urine collection from baseline to end of treatment period
Urinary potassium | 12 weeks
  Change in urinary potassium levels (mmol per liter) in one 24h urine collection from baseline to end of treatment period

OTHER OUTCOMES:
Safety outcome - Adverse events | 12 weeks
  Total number of adverse events from baseline to end of treatment
Safety outcome - Electrocardiogram | 12 weeks
  Number of adverse events related to changes in the electrocardiogram (e.g. QTc prolongation) from baseline to end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No